CLINICAL TRIAL: NCT06866041
Title: Biological Pathways and Next-Generation Imaging Features Predicting Prostate Cancer Progression in Active Surveillance
Brief Title: Biological Markers and Advanced Imaging for Prostate Cancer Progression in Active Surveillance
Acronym: PSMA-AS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giorgio Gandaglia, Medical Doctor, Università Vita-Salute San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSMA-AS
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Low-Risk Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): All patients with low-risk prostate cancer (ISUP Grade Group 1) eligible for active surveillance will undergo:
  * PSMA-PET/MRI → Evaluation of intraprostatic PSMA expression (SUVmax, PRIMARY-likert score).
  * Whole Exome Sequencing (WES) → Genomic analysis of diagnostic biopsies. Multiplex Immunohistochemistry (IHC) → Study of biomarkers on diagnostic biopsies.
  Confirmation biopsy one year after diagnosis, according to international guidelines.
  Interventions: Procedure: mpMRI-targeted confirmatory biopsy

INTERVENTIONS:
Procedure: mpMRI-targeted confirmatory biopsy — mpMRI-targeted confirmatory biopsy after one year from the diagnosis, according to the international guidelines
  Other Names: 18F-PSMA PET/MRI; WES and spatial transcriptomics on the diagnostic biopsy specimens; Multiplex immunohistochemistry on the diagnostic biopsy specimens

SUMMARY:
This study aims to identify patients with low-risk prostate cancer (ISUP Grade Group 1) eligible for active surveillance who are at higher risk of upgrading to ISUP Grade Group 2 or higher at confirmatory biopsy one year after diagnosis. Patients with low-risk ISUP GG1 tumors will be selected and undergo:

* PSMA PET with calculation of SUVmax and PRIMARY-Likert score
* Whole Exome Sequencing (WES) analysis on diagnostic prostate biopsies
* Immunohistochemistry on diagnostic prostate biopsies
* Confirmatory biopsy one year after diagnosis, as recommended by international guidelines This prospective, monocentric, single-arm interventional study will assess the predictive accuracy of a multivariable model integrating next-generation imaging and molecular biomarkers to improve risk stratification in active surveillance patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven low-risk PCa (PSA ≤10 ng/ml; clinical stage ≤T2a, and biopsy ISUP GG 1)
* Non-metastatic status at study inclusion (patient enrollment).
* No prior or concomitant androgen deprivation therapy
* Ability to understand a written informed consent and willingness to sign it.

Exclusion Criteria:

* Unable to tolerate a PSMA-PET scan
* Unwillingness to be managed with AS
* Receipt of neoadjuvant or curative-intent therapies
* Pacemaker
* Inability to obtain the FFPE prostate biopsy specimens from the initial biopsy

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-05-07 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Discriminative Ability of a Multivariable Model in Predicting Prostate Cancer Upgrading in Low-Risk Patients Under Active Surveillance" | Baseline diagnostic biopsy and 12 months after diagnosis (when the confirmatory biopsy will be performed)
  To determine the discriminative ability of the multivariable model, quantified using the concordance index (c-index), to predict prostate cancer upgrading in low-risk PCa patients managed with active surveillance (AS).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy